CLINICAL TRIAL: NCT00959452
Title: Follow up of Patients Treated With Cognitive Behavioural Therapy at Clinic for Hypochondriacs, Haraldsplass Deaconal Hospital, From 1997 to 2007
Brief Title: Follow up of Patients Treated With Cognitive Behavioural Therapy for Hypochondria From 1997 to 2007
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Ingvard Wilhelmsen, Professor emeritus, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17242
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Hypochondriasis
Keywords: Hypochondria; Cognitive behavioural therapy; Long term follow-up; Psychosomatics; Psychotherapy
MeSH Terms: conditions — Hypochondriasis | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychotherapy (Experimental)
  Interventions: Behavioral: Cognitive behavioural therapy

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — 16 sessions vs 5 sessions of cognitive behavioural therapy
  Other Names: Cognitive therapy

SUMMARY:
Research has shown that cognitive behavioural therapy is effective in treating hypochondria. However, no studies have examined the long term effect. The investigators have followed 56 patients treated for hypochondria between 1997 and 2001 and the investigators are now doing a 10 year follow-up (Part I). In another part of the study (Part II) the investigators compare the effect of 16 sessions vs. 5 sessions, with a follow-up period of at least 2 years. The investigators hypothesis is that the initial 1 year improvement will be sustained and that 5 sessions will yield the same results as 16 sessions.

DETAILED DESCRIPTION:
The follow-up includes a telephone interview by independent researcher and the patients fill in the following questionnaires:

Whiteley Index (measures health anxiety), VAS-scales for health anxiety, worrying about symptoms and body checking, SF-36 (health related quality of life), Giessen Subjective Complaints List, Spielberger Trait and State Anxiety Scale Beck Depression Inventory, Eysenck Personality Questionnaire, General Health Questionnaire (GHQ 28), Somatic Amplification Scale,

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling ICD-10 criteria for hypochondriacal disorder

Exclusion Criteria:

* Unwillingness to participate
* Substance abuse
* Serious psychological (f.inst. psychosis, major depression) or somatic (f.inst. cancer) disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 1997-01; Primary Completion 2010-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Level of health anxiety | 10 years follow up

SECONDARY OUTCOMES:
Health related quality of life | 10 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ingvard Wilhelmsen, PhD, Principal Investigator — University of Bergen
Locations (1):
- Haraldsplass Deaconal Hospital, Bergen, Norway

REFERENCES:
- [Result] Veddegjaerde KE, Sivertsen B, Wilhelmsen I, Skogen JC. Confirmatory factor analysis and item response theory analysis of the Whiteley Index. Results from a large population based study in Norway. The Hordaland Health Study (HUSK). J Psychosom Res. 2014 Sep;77(3):213-8. doi: 10.1016/j.jpsychores.2014.06.011. Epub 2014 Jun 28. PMID 25149031
- [Result] Veddegjaerde KF, Sivertsen B, Skogen JC, Smith ORF, Wilhelmsen I. Long-term effect of cognitive-behavioural therapy in patients with Hypochondriacal Disorder. BJPsych Open. 2020 Apr 29;6(3):e42. doi: 10.1192/bjo.2020.22. PMID 32345417